CLINICAL TRIAL: NCT00378482
Title: A Rollover Protocol For Patients Who Received Tremelimumab (CP-675,206 ) In Other Protocols
Brief Title: A Rollover Study for Patients Who Received Tremelimumab in Other Protocols, to Allow the Patients Access to Tremelimumab Until This Agent Becomes Commercially Available or Development is Discontinued.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: D4881C00024; D4881C00024 (A3671024) (Other: AZ study code); 2008-000989-23 (EudraCT Number)
Record Dates: First submitted 2006-09-19; First posted 2006-09-20 (Estimated); Results first posted 2021-05-28 (Actual); Last update posted 2024-08-22 (Actual); Status verified 2024-08

CONDITIONS: Colorectal Neoplasms; Melanoma; Prostatic Neoplasms; Renal Cell Carcinoma; Neoplasms; Patients Who Have/Have Had Melanoma and Other Tumors
Keywords: Melanoma and other tumors
MeSH Terms: conditions — Colorectal Neoplasms; Melanoma; Prostatic Neoplasms; Carcinoma, Renal Cell; Neoplasms | interventions — tremelimumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): Drug: CP-675,206 (Tremelimumab)
  Interventions: Drug: CP-675,206 (Tremelimumab)

INTERVENTIONS:
Drug: CP-675,206 (Tremelimumab) — 15 mg/kg IV every 3 months as long as required
  Other Names: anti-CTLA4 human monoclonal antibody

SUMMARY:
This study is intended to provide access to tremelimumab for patients who have previously received tremelimumab in a clinical trial.

ELIGIBILITY:
Inclusion Criteria:

* The subject must have already received tremelimumab in another protocol
* Females of childbearing potential must agree to practice a form of effective contraception for 12 months following any dose of study drug. The definition of effective contraception will be based on the judgement of the investigator.
* Subject must be willing and able to provide written informed consent and to comply with scheduled visits and other trial procedures

Exclusion Criteria:

* None

Ages: 18 Years to 130 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2007-03-05 (Actual); Primary Completion 2023-10-27 (Actual); Study Completion 2023-10-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: AstraZeneca AstraZeneca, Study Director — AstraZeneca; Peter Langmuir, Dir.Medic.Science, Study Director — AstraZeneca
Locations (6):
- United States (5):
  - Research Site, Los Angeles, California
  - Research Site, Tampa, Florida
  - Research Site, Ann Arbor, Michigan
  - Research Site, New York, New York
  - Research Site, Houston, Texas
- Research Site, Newecastle Upon Tyne, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal. All request will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure
Supporting Information: Study Protocol, SAP
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the de-identified individual patient-level data in an approved sponsored tool . Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home

REFERENCES:
- See also: Redacted SAP — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D4881C00024&attachmentIdentifier=5ab57894-fa70-4755-a7d3-41e1d89888d7&fileName=D4881C00024_SAP_redacted.pdf&versionIdentifier=
- See also: Redacted CSP — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D4881C00024&attachmentIdentifier=098db55e-fbbb-4d63-abe9-e79e302970cc&fileName=D4881C00024-csp_redacted.pdf&versionIdentifier=
- See also: CSR Synopsis — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D4881C00024&attachmentIdentifier=ae993f6e-251e-4dce-ac8a-35e07d7aa8ff&fileName=d4881c00024-clinical-study-report_synopsis.pdf&versionIdentifier=

RESULTS

PARTICIPANT FLOW:
Recruitment Details: First subject enrolled: 05 Mar 2007; Data Cut-off: 18 Jun 2020. This was a multicenter study conducted at 11 study centers in 3 countries (the United Kingdom, the United States of America and Italy).
Pre-assignment Details: Total Consented/screened 38 subjects (1 of which was dead before enter any treatment), so total entered treatment 37 subjects. Subjects were assigned to treatment if they met all inclusion. 32 subjects withdrawn from this study. 6 subjects completed the study.
  Final Efficacy/Safety analysis 37 subjects.
Groups:
- Tremelimumab 15mg/kg: All Patients
Period: Overall Study
Arm/Group | Tremelimumab 15mg/kg
Started (37) | 37
Completed (6) | 6
Not Completed | 31
Not completed — Lost to Follow-up | 1
Not completed — Lack of Efficacy | 8
Not completed — Subject or physician decision, or subject relocation to another city or region. | 9
Not completed — Withdrawal by Subject | 4
Not completed — Adverse Event | 9

BASELINE CHARACTERISTICS:
Population: One participant received no study medication and was excluded from data analysis
Arm/Group | Tremelimumab 15mg/kg
Number analyzed (Participants) | 37
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 24
  >=65 years | 13
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 26
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 37
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Safety Endpoints: Serious Adverse Events to Tremelimumab.
Time Frame: Following the first dose, until at least 90 days since the previous dose of tremelimumab or at least 28 days since any study-related procedures. Actual median study duration was 2.2 years.
Population: 37 Participants received study treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Tremelimumab 15mg/kg
Number analyzed (Participants) | 37
Participants
  Number of Participants with SAE to tremelimumab | 4
  Number of Participants with no SAE to tremelimumab | 33

2. Primary Outcome: Safety Endpoints: Grade 3 or 4 Tremelimumab-related Adverse Events to Tremelimumab.
Time Frame: as for outcome 1
Population: 37 Participants received study treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Tremelimumab 15mg/kg
Number analyzed (Participants) | 37
Participants
  Number of participants with Grade 3 or 4 tremelimumab-related adverse events to tremelimumab | 4
  Number of participants with no Grade 3 or 4 tremelimumab-related adverse events to tremelimumab | 33

3. Primary Outcome: Safety Endpoints: Hypersensitivity Reactions to Tremelimumab.
Time Frame: as for outcome 1
Population: 37 Participants received study treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Tremelimumab 15mg/kg
Number analyzed (Participants) | 37
Participants
  Number of participants with Hypersensitivity reactions to tremelimumab | 6
  Number of participants with no Hypersensitivity reactions to tremelimumab | 31

4. Primary Outcome: Efficacy Endpoints: Tumor Status: Alive With Disease (AWD) or no Evidence of Disease (NED)
Time Frame: as for outcome 1
Population: Treated patients with response assessed
Measure: Count of Participants; unit: Participants
Arm/Group | Tremelimumab 15mg/kg
Number analyzed (Participants) | 37
Participants
  No evidence of disease | 19
  Evidence of disease | 17
  Indeterminate | 1

5. Primary Outcome: Efficacy Endpoints: Survival
Time Frame: as for outcome 1
Population: Treated patients with response assessed
Measure: Count of Participants; unit: Participants
Arm/Group | Tremelimumab 15mg/kg
Number analyzed (Participants) | 37
Participants
  Death | 10
  Censored | 27

6. Secondary Outcome: Disease Free Survival
Description: Time from the first dose of study drug to the earliest date of evidence of disease (based on tumor status assessment) or death, whichever occurred first
Time Frame: as for outcome 1
Population: Treated patients
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Tremelimumab 15mg/kg
Number analyzed (Participants) | 37
Days | 3.0 [2.9 to 11.8]

ADVERSE EVENTS:
Time Frame: 13 years, 3 months
Arm/Group | Tremelimumab 15mg/kg
All-Cause Mortality (participants affected / at risk) | 11/37
Serious Adverse Events (participants affected / at risk) | 4/37
Other Adverse Events (participants affected / at risk) | 5/37
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tremelimumab 15mg/kg (N=37)
Diarrhea (Gastrointestinal disorders) | 1 (1)
Medical Device Complication (General disorders) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 1 (1)
Sepsis (Infections and infestations) | 1 (1)
Urinary Tract Infection (Infections and infestations) | 1 (1)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Pulmonary Granuloma (Respiratory, thoracic and mediastinal disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tremelimumab 15mg/kg (N=37)
Rash (Skin and subcutaneous tissue disorders) | 4 (12)
Pruritus (Skin and subcutaneous tissue disorders) | 3 (3)
Hypothyroidism (Endocrine disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor can review results communications prior to public release and can embargo regarding trial results for up to six (6) months from the time submitted to the sponsor for review. All reasonable comments made by the sponsor in relation to the publication will be incorporated into the publication. PI shall not unreasonable withhold or delay its consent to a request from the sponsor for an exceptional additional delay if in the reasonable opinion of the sponsor.

DOCUMENTS (2):
  • Study Protocol (2019-12-26): https://cdn.clinicaltrials.gov/large-docs/82/NCT00378482/Prot_000.pdf
  • Statistical Analysis Plan (2020-02-17): https://cdn.clinicaltrials.gov/large-docs/82/NCT00378482/SAP_001.pdf